CLINICAL TRIAL: NCT01836185
Title: Pharmacokinetics of Evacetrapib (LY2484595) in Subjects With Hepatic Impairment
Brief Title: A Study of Evacetrapib (LY2484595) in Participants With Hepatic (Liver) Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 14621; I1V-MC-EIAS (Other: Eli Lilly and Company)
Record Dates: First submitted 2013-04-17; First posted 2013-04-19 (Estimated); Results first posted 2018-10-12 (Actual); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Hepatic Insufficiency
MeSH Terms: conditions — Hepatic Insufficiency | interventions — evacetrapib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Evacetrapib (Healthy) (Experimental): Group 1: 130 milligrams (mg) evacetrapib administered once, orally, to participants with normal hepatic function
  Interventions: Drug: Evacetrapib
- Evacetrapib (Hepatic, Mild) (Experimental): Group 2: 130 mg evacetrapib administered once, orally, to participants with mild hepatic impairment
  Interventions: Drug: Evacetrapib
- Evacetrapib (Hepatic, Moderate) (Experimental): Group 3: 130 mg evacetrapib administered once, orally, to participants with moderate hepatic impairment
  Interventions: Drug: Evacetrapib
- Evacetrapib (Hepatic, Severe) (Experimental): Group 4: 130 mg evacetrapib administered once, orally, to participants with severe hepatic impairment
  Interventions: Drug: Evacetrapib

INTERVENTIONS:
Drug: Evacetrapib
  Other Names: LY2484595

SUMMARY:
The purpose of this study is to measure how much of the drug gets into the bloodstream and how long it takes the body to remove it when given to participants with hepatic (liver) impairment compared to participants with normal hepatic function. Information about any side effects that may occur will also be collected. This study will last approximately 28 days, not including screening.

ELIGIBILITY:
Inclusion Criteria:

* Participants have given written informed consent approved by the ethical review board (ERB) governing the site
* Female participants should be of non-childbearing potential
* Have a body mass index (BMI) of 18 to 40 kilograms per square meter (kg/m^2)
* Healthy participants have normal hepatic function as determined by medical history, physical examination, and other screening procedures
* Individuals with hepatic impairment classified as Child-Pugh score A, B, or C (mild, moderate, or severe impairment)

Exclusion Criteria:

* Has had esophagus variceal bleeding within 3 months of check-in
* Have the need to take medications that may interfere with how the liver removes the drug
* Have evidence of cancer in the liver
* Consumes excessively large amounts of drinks with caffeine or alcohol

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-04; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- United States (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miami, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orlando, Florida

RESULTS

PARTICIPANT FLOW:
Groups:
- Evacetrapib (Healthy): Group 1: 130 milligrams (mg) evacetrapib administered once, orally as a tablet to participants with normal hepatic function
- Evacetrapib (Hepatic, Mild): Group 2: 130 mg evacetrapib administered once, orally as a tablet to participants with mild hepatic impairment
- Evacetrapib (Hepatic, Moderate): Group 3: 130 mg evacetrapib administered once, orally as a tablet to participants with moderate hepatic impairment
- Evacetrapib (Hepatic, Severe): Group 4: 130 mg evacetrapib administered once, orally as a tablet to participants with severe hepatic impairment
Period: Overall Study
Arm/Group | Evacetrapib (Healthy) | Evacetrapib (Hepatic, Mild) | Evacetrapib (Hepatic, Moderate) | Evacetrapib (Hepatic, Severe)
Started | 10 | 8 | 8 | 6
Received Single Dose of Study Treatment | 10 | 8 | 8 | 6
Completed | 10 | 8 | 8 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Evacetrapib (Healthy) | Evacetrapib (Hepatic, Mild) | Evacetrapib (Hepatic, Moderate) | Evacetrapib (Hepatic, Severe) | Total
Number analyzed (Participants) | 10 | 8 | 8 | 6 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.4 (8.6) | 54.1 (2.9) | 58.6 (9.6) | 57.8 (4.7) | 56.0 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 2 | 1 | 11
  Male | 6 | 4 | 6 | 5 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 2 | 4 | 3 | 17
  Not Hispanic or Latino | 2 | 6 | 4 | 3 | 15
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 0 | 2
  White | 9 | 6 | 8 | 6 | 29
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 8 | 8 | 6 | 32

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve From Time Zero to Time Tlast (AUC0-tlast) of Evacetrapib
Description: tlast is defined as the last time point with a measurable concentration of Evacetrapib.
Time Frame: Predose on Day 1, and 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 120, 168, 216, 264, 312, and 336 hours after the Day 1 dose
Population: Participants who received at least 1 dose of study drug and had evaluable PK (AUC0-tlast) data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour per milliliter (ng*h/mL)
Groups:
- Evacetrapib (Healthy): Group 1: 130 mg evacetrapib administered once, orally as a tablet to participants with normal hepatic function
Arm/Group | Evacetrapib (Healthy) | Evacetrapib (Hepatic, Mild) | Evacetrapib (Hepatic, Moderate) | Evacetrapib (Hepatic, Severe)
Number analyzed (Participants) | 10 | 8 | 8 | 6
nanograms*hour per milliliter (ng*h/mL) | 10700 (50) | 10500 (84) | 13200 (49) | 15800 (62)

2. Primary Outcome: PK: Maximum Observed Concentration (Cmax) of Evacetrapib
Time Frame: Predose on Day 1, and 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 120, 168, 216, 264, 312, and 336 hours after the Day 1 dose
Population: Participants who received at least 1 dose of study drug and had evaluable PK (Cmax) data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Evacetrapib (Healthy) | Evacetrapib (Hepatic, Mild) | Evacetrapib (Hepatic, Moderate) | Evacetrapib (Hepatic, Severe)
Number analyzed (Participants) | 10 | 8 | 8 | 6
ng/mL | 605 (98) | 609 (144) | 591 (58) | 478 (51)

3. Primary Outcome: PK: Time of Maximum Observed Drug Concentration (Tmax) of Evacetrapib
Time Frame: Predose on Day 1, and 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 120, 168, 216, 264, 312, and 336 hours after the Day 1 dose
Population: Participants who received at least one dose of study drug and had evaluable PK data.
Measure: Mean (Full Range); unit: h
Arm/Group | Evacetrapib (Healthy) | Evacetrapib (Hepatic, Mild) | Evacetrapib (Hepatic, Moderate) | Evacetrapib (Hepatic, Severe)
Number analyzed (Participants) | 10 | 8 | 8 | 6
h | 3 [2 to 6] | 3 [1 to 4] | 3 [2 to 4] | 3 [2 to 6]

ADVERSE EVENTS:
Time Frame: Randomization to study completion (Up To 41 Days)
Groups:
- Evacetrapib (Hepatic, Moderate): Group 3: 130 mg evacetrapib administered once, orally, as a tablet to participants with moderate hepatic impairment
Arm/Group | Evacetrapib (Healthy) | Evacetrapib (Hepatic, Mild) | Evacetrapib (Hepatic, Moderate) | Evacetrapib (Hepatic, Severe)
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/8 | 0/8 | 0/6
Other Adverse Events (participants affected / at risk) | 2/10 | 4/8 | 3/8 | 3/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Evacetrapib (Healthy) (N=10) | Evacetrapib (Hepatic, Mild) (N=8) | Evacetrapib (Hepatic, Moderate) (N=8) | Evacetrapib (Hepatic, Severe) (N=6)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Piloerection (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days